CLINICAL TRIAL: NCT02666261
Title: A Non-interventional Study on the Epidemiology and Testing of HER2 in Breast Cancer in Germany
Brief Title: A Study on the Epidemiology and Testing of Human Epidermal Growth Factor-Receptor 2 (HER2) in Breast Cancer in Germany
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML29763
Record Dates: First submitted 2016-01-11; First posted 2016-01-28 (Estimated); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Breast Cancer Pathology Samples: Data on the epidemiology and HER2 testing of breast cancer will be collected from pathology routine diagnostics.

SUMMARY:
This non-interventional study will collect data from routine diagnostics on HER2 testing of breast cancer in Germany.

ELIGIBILITY:
Inclusion Criteria:

* Samples derived from men and women of age greater than or equal to (>/=) 18 years
* Samples derived from participants with any stage of histologically confirmed invasive breast cancer with HER2 diagnostics performed within routine (histo-)pathological workup or
* (Histo-)Pathological work-up of the tumor sample as at or after start of this study
* Available information on the year of birth of the participant
* No pre-selection of tumor samples is allowed. Tumor samples have to be documented consecutively in the order of their (histo-)pathological work-up.

Exclusion Criteria:

* Sample derived from participants with any stage of breast cancer with no HER2 diagnostics performed at the time of routine (histo-)pathological work-up.
* Samples derived prior to the start of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer tissue samples from participants in Germany
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2016-03-04 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Number of HER2 Positive Samples | 1 day (this is a single time point study)

SECONDARY OUTCOMES:
Number of HER2 Positive Samples by Carcinoma Subtype (No Special Type\Ductal, Lobular, Other Special Type) | 1 day (this is a single time point study)
Number of HER2 Positive Samples by Sample Extraction (Biopsy versus Resectate) | 1 day (this is a single time point study)
Number of HER2 Positive Samples by Tumor-Node-Metastasis (TNM) Classification | 1 day (this is a single time point study)
Number of HER2 Positive Samples by Sample Source (Primary Tumor, Local Lymph Nodes, Metastasis) | 1 day (this is a single time point study)
Number of HER2 Positive Samples by Applied Method of Tissue Fixation | 1 day (this is a single time point study)
Number of HER2 Positive Samples by Testing Platform | 1 day (this is a single time point study)
Number of HER2 Positive Samples by Automation of Testing | 1 day (this is a single time point study)
Number of HER2 Positive Samples by Antibody Clone Antibody or Test Certification | 1 day (this is a single time point study)
Number of HER2 Positive Samples by Scoring Algorithm | 1 day (this is a single time point study)
Number of HER2 Positive Samples by Round Robin Tests | 1 day (this is a single time point study)
Number of HER2 Positive Samples by Institute's Accreditation | 1 day (this is a single time point study)
Number of HER2 Positive Samples by Institute's Certification | 1 day (this is a single time point study)
Number of HER2 Positive Samples by Tumor Grading | 1 day (this is a single time point study)
Number of HER2 Positive Samples by Participant Age | 1 day (this is a single time point study)
Number of HER2 Positive Samples by Hormone Receptor Status | 1 day (this is a single time point study)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (64):
- Germany (64):
  - Klinikum Augsburg; Institut für Pathologie, Augsburg
  - Sozialstiftung Bamberg; Institut für Pathologie, Bamberg
  - Klinikum Bayreuth, Bayreuth
  - Institut für Pathologie, Zytologie & Molekularpathologie in Bergisch Gladbach, Bergisch Gladbach
  - Gemeinschaftspraxis für Pathologie Stefan Berger, Jörg Linke und Ellen Fietze, Berlin
  - Vivantes Klinikum Neukölln; Fachbereich Pathologie, Berlin
  - HELIOS Klinikum Emil von Behring Klinik f.Pneumologie Onkologie u.Infektiologie, Berlin
  - Gemeinschaftspraxis; Institut für Pathologie am Evangelischen Waldkrankenhaus, Berlin - Spandau
  - Praxis am St. Agnes-Hospital Bocholt, Bocholt
  - Institut für Pathologie und Zytologie an der Augusta-Kranken-Anstalt, Bochum
  - Universitätsklinikum Bonn; Zentrum für Pathologie Pathologisches Institut, Bonn
  - Klinikum Coburg GmbH - Institut für Pathologie, Coburg
  - Institut f. Pathologie, der Univers. Köln, Cologne
  - Kliniken der Stadt Köln gGmbH Krankenhaus Merheim, Cologne
  - Städtisches Klinikum Dessau; Institut für Pathologie, Dessau
  - Gemeinschaftspraxis für Pathologie Dr. Dykgers, Dr. Langwieder, Dr. Rees, Dortmund
  - Städtisches Klinikum Dresden; Institut für Pathologie "Georg Schmorl" (Friedrichstadt), Dresden
  - Evangelisches Krankenhaus BETHESDA zu Duisburg GmbH; Institut für Pathologie, Duisburg
  - Krankenhaus Düren gem. GmbH; Institut und Praxisgemeinschaft für Pathologie, Düren
  - Universitätsklinikum Erlangen; Pathologisches Institut, Erlangen
  - OptiPath Gemeinschaftspraxis für Pathologie, Frankfurt
  - Universitätsklinikum Freiburg Institut f.Pathologie, Freiburg im Breisgau
  - Pathologische Institut Friedrichshafen/Bodensee (Gemeinschaftspraxis für Pathologie und Zytologie), Friedrichshafen
  - Klinik am Eichert; Institut für Pathologie, Göppingen
  - Universitätsklinikum Göttingen, Institut für Pathologie, Göttingen
  - Institut für Pathologie, MVZ am Lukaskrankenhaus, Grevenbroich
  - Klinikum Oberberg; Pathologisches Institut Kreiskrankenhaus Gummersbach, Gummersbach
  - Pathologisches Institut am Allg. KH Stadt Hagen; Stambolis, Wolf von Rhüden, Ruwe, Hagen
  - Universitätsklinikum Halle (Saale), Institut für Pathologie, Halle
  - Kath. Marienkrankenhaus gGmbH, Hamburg
  - Fachärzte Dres Tiemann & Schulte Partnerschaft; Institut für Hämatopathologie Hamburg, Hamburg
  - Gemeinschaftspraxis für Pathologie Hamm, Dres. Diebold/Niemann, Hamm
  - Gemeinschaftspraxis Dr. Hartmut Fitz, Dr. Sebastian Blasius und PD Dr. Christian August, Hanau
  - Dres. Wolfgang Beschow Eckehardt Kupsch Herbert Radner u.w., Hanover
  - Medizinische Hochschule Hannover, Klinik für Frauenheilkunde und Geburtshilfe, Hanover
  - Pathologisches Institut, Heidelberg
  - Institut für Pathologie Hildesheim, Hildesheim
  - Gemeinschaftspraxis für Pathologie Ingolstadt Dr. König, Dr. Popp, Prof. Dr. Adam, Ingolstadt
  - Universitätsklinikum Jena; Institut für Pathologie, Jena
  - Städtisches Klinikum Karlsruhe gGmbH; Pathologisches Institut, Karlsruhe
  - Institut Für Pathologie Nordhessen, Kassel
  - Institut für Pathologie Kassel, Kassel
  - Institut für Pathologie, Universitäsklinikum Schleswig-Holstein, Kiel
  - Klinikum Konstanz gGmbH, Institut und Praxis für Pathologie, Konstanz
  - Gemeinschaftspraxis für Pathologie Lübeck; Turzynski, Lebeau, Gocht, Leuenroth, Lübeck
  - Universitätsklinikum Magdeburg; Institut für Pathologie und Neuropathologie, Magdeburg
  - Klinikum Magdeburg GmbH, Magdeburg
  - Klinikum Mannheim; Pathologisches Institut, Mannheim
  - Institut für Pathologie, Mühlhausen
  - Pathologie München-Nord, München
  - Institut für Pathologie der Universität Münster, Albert Schweitzer Campus, Gebäude D17, Münster
  - Institut für Pathologie am Clemenshospital Münster, Münster
  - Dietrich Bonhoeffer Kliniken Neubrandenburg, Institut für Pathologie, Neubrandenburg
  - Zentrum für Pathologie, Zytologie und Molekularpathologie Neuss, Neuss
  - Evangelisches Krankenhaus Oberhausen GmbH, Institut f.Pathologie, Oberhausen
  - Pathocom - Gemeinschaftspraxis Bischofsstraße Osnabrück, Osnabrück
  - Pathologisches Institut Recklinghausen, Recklinghausen
  - Klinikum am Steinenberg / Ermstalklinik, Reutlingen
  - Diakoniekrankenhaus Institut f.Pathologie, Rotenburg (Wümme)
  - Leopoldina Krankenhaus der Stadt Schweinfurt GmbH; Pathologie, Schweinfurt
  - HELIOS Klinikum Schwerin; Frauenklinik, Schwerin
  - Gemeinschaftspraxis PD Dr.med. Meinald Schultz und Dr.med. Petra Lüders, Stendal
  - Robert-Bosch-Krankenhaus; Pathologisches Institut, Stuttgart
  - Gemeinschaftspraxis für Pathologie Weiden; am Klinikum Weiden; Giedl, Stelter und Meier, Weiden